CLINICAL TRIAL: NCT01206608
Title: A Randomized, Double-Blind, Active-Control Study to Evaluate the Safety and Efficacy of a Single Local Administration of SKY0402 for Prolonged Postoperative Analgesia in Subjects Undergoing Augmentation Mammoplasty
Brief Title: Evaluation of the Safety and Efficacy of a Single Dose of SKY0402 in Subjects Undergoing Augmentation Mammoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402-C-210
Record Dates: First submitted 2010-09-19; First posted 2010-09-22 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
Keywords: Breast augmentation; Pain; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-dose SKY0402 + bupivacaine HCl (Active Comparator): Marcaine with epinephrine 1:200,000 is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402
  Interventions: Drug: SKY0402 + bupivacaine HCl
- Mid-dose SKY0402 + bupivacaine HCl (Active Comparator): Marcaine with epinephrine 1:200,000 is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402
  Interventions: Drug: Mid-dose SKY0402 + bupivacaine HCl

INTERVENTIONS:
Drug: SKY0402 + bupivacaine HCl — Low-dose SKY0402 administered locally into one breast pocket and 75 mg bupivacaine HCl administered locally into the other breast pocket
  Arms: Low-dose SKY0402 + bupivacaine HCl
Drug: Mid-dose SKY0402 + bupivacaine HCl — Mid-dose SKY0402 administered locally into one breast pocket and 75 mg bupivacaine HCl administered locally into the other breast pocket
  Arms: Mid-dose SKY0402 + bupivacaine HCl

SUMMARY:
The primary objective of this study was to demonstrate the superiority of SKY0402 over conventional, commercially-available bupivacaine HCl with respect to the duration of the analgesic effect achieved by a single local administration of the study drug.

DETAILED DESCRIPTION:
This was a Phase 2, parallel-group, active-control, randomized, double-blind study conducted to evaluate a single local administration of low dose or high dose of SKY0402 compared with 75 mg of bupivacaine HCl (i.e., Marcaine® 0.5%) in women undergoing bilateral, cosmetic, sub-muscular, augmentation mammoplasty under general anesthesia. Each subject was to serve as her own control.

A total of 40 subjects were randomized in a 1:1 ratio to receive one of the following regimens:

* Low-dose SKY0402 in one side and Marcaine 75 mg in the contralateral side.
* Mid-dose SKY0402 in one side and Marcaine 75 mg in the contralateral side.

Study drug was administered locally into the breast implant pocket at the end of surgery. After surgery, subjects were to receive standard treatment with acetaminophen 1000 mg three times daily and rescue analgesia with immediate-release oxycodone, as needed, for breakthrough pain.

Assessments of postoperative pain were conducted through 96 hours. Safety assessments were conducted including monitoring of local and systemic adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

Subjects who met all of the following criteria were eligible for inclusion in the study:

1. Women, 18-40 years of age at the Screening Visit.
2. Postmenopausal, surgically sterile, or willing to use an acceptable means of contraception for at least 30 days after surgery including any of the following: hormonal contraceptives (e.g., oral, injectable, implantable starting at least 30 days before study drug administration), effective double-barrier methods (e.g., condoms with spermicide), intrauterine device, lifestyle with a personal choice of abstinence, nonheterosexual lifestyle, or a strictly monogamous relationship with a partner who has had a vasectomy.
3. Scheduled to undergo primary, bilateral, sub-muscular, augmentation mammoplasty under general anesthesia.
4. American Society of Anesthesiology (ASA) Physical Class 1-3.
5. Able and willing to comply with all study visits and procedures.
6. Able to speak, read, and understand the language of the ICF, study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.
7. Willing and capable of providing written informed consent.

Exclusion Criteria:

* Subjects were not eligible for the study if they met any of the following criteria:

  1. Pregnancy, nursing, or planning to become pregnant during the study or within one month after study drug administration.
  2. Body weight less than 50 kilograms.
  3. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics or to opioid medication.
  4. Administration of an investigational product within 30 days or 5 elimination half-lives of such investigational product, whichever was longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
  5. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
  6. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
  7. Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicated an increased vulnerability to study drugs and procedures, and exposed the subject to an unreasonable risk as a result of participating in this clinical trial (e.g., severe hepatic insufficiency, hypotension, heart block, or severely impaired cardiac function).

     In addition, the subject was ineligible to receive study drug if she met the following criterion during surgery:
  8. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postoperative course.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, ACNP, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- Associates for Plastic Surgery, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-dose SKY0402 + Bupivacaine HCl | Mid-dose SKY0402 + Bupivacaine HCl
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose SKY0402 + Bupivacaine HCl | Mid-dose SKY0402 + Bupivacaine HCl | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (7) | 28.4 (6) | 29.6 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) at Rest (NRS-R) and With Activity (NRS-A) Pain Intensity Scores
Description: Assessments of postoperative pain were conducted through 96 hours and included pain intensity at rest (NRS-R) and with activity (NRS-A). The prescribed activity was to consist of raising the arm, in full extension at the elbow and wrist, to a position parallel with the axis of the torso. Pain intensity was scored on an 11-point scale, where 0 = no pain and 10 = worst possible pain.
Time Frame: Through 96 hours postdose
Measure: Mean (Standard Deviation); unit: Units on a scale*hours
Groups:
- Low-dose SKY0402 (150mg) + Bupivacaine HCl; Mid-dose SKY0402 (300mg)+ Bupivacaine HCl: Marcaine with epinephrine 1:200,000 is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402. A single dose of 150mg SKY0402 administration via local infiltration.
Arm/Group | Low-dose SKY0402 (150mg) + Bupivacaine HCl | Mid-dose SKY0402 (300mg)+ Bupivacaine HCl
Number analyzed (Participants) | 20 | 20
Units on a scale*hours | 340.7 (141.6) | 293.4 (194.2)

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were monitored through Day 8 and serious adverse events through Day 30.
Time Frame: Through 30 days postdose
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Low-dose SKY0402 + Bupivacaine HCl | Mid-dose SKY0402 + Bupivacaine HCl
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 19/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-dose SKY0402 + Bupivacaine HCl (N=20) | Mid-dose SKY0402 + Bupivacaine HCl (N=20)
Postprocedural hematoma (Injury, poisoning and procedural complications) | 0 | 1 — Occurred locally in the breast exposed to bupivacaine only
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low-dose SKY0402 + Bupivacaine HCl (N=20) | Mid-dose SKY0402 + Bupivacaine HCl (N=20)
Tachycardia (Cardiac disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 16 | 13
Vomiting (Gastrointestinal disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No